CLINICAL TRIAL: NCT06185907
Title: In-hospital Outcomes of Older Patients With Gastric Cancer and Their Risk Factors: Large Comprehensive Institution-based Study
Brief Title: In-hospital Outcomes of Older Patients With Gastric Cancer and Their Risk Factors
Acronym: GGC-01
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, lei huang, Principal investigator, Ruijin Hospital
Other Study IDs: GGC-01
Record Dates: First submitted 2023-11-27; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric gastric cancer patients
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — We referr to resection as that performed in our hospital, and history of major abdominal surgery as interventional surgical procedures in the abdomen with therapeutic intent (e.g., resection) prior to the first hospitalization in our hospital.

SUMMARY:
The investigators plan to analyze the data of patients with gastric cancer (GC) consecutively hospitalized in Ruijin Hospital, a large tertiary center in China, comprehensively describe the characteristics of GC patients ≥65 years, and assesse their in-hospital outcomes regarding duration, fee, and death. Factors associated with the in-hospital outcomes will be further comprehensively explored.

ELIGIBILITY:
Inclusion Criteria:

* Older gastric cancer (GC) patients
* With primary malignancies of the stomach (International Classification of Diseases for Oncology, Third Edition [ICD-O-3] topology code: C16)
* ≥65 years

Exclusion Criteria:

* With benign, premalignant, or in situ tumors
* With cancers originating from non-stomach sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males takes up 74% of the entire population, whose median age is 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 3238 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 1 month
  Mortality during first and all hospitalizations
Cost | Up to 1 month
  Costs during first and all hospitalizations
Duration of stay | Up to 1 month
  Duration of stay during first and all hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China